CLINICAL TRIAL: NCT05568069
Title: Using Cardiovascular Magnetic Resonance Identified Scar as the Benchmark Risk Indication Tool for Implantable Cardioverter Defibrillators in Patients With Non-Ischemic Cardiomyopathy and Severe Systolic Heart Failure
Brief Title: RCT of Implantable Defibrillators in Patients With Non Ischemic Cardiomyopathy, Scar and Severe Systolic Heart Failure
Acronym: BRITISH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: British Heart Foundation (Other); University of Southampton (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RHMCAR0581
Record Dates: First submitted 2022-09-27; First posted 2022-10-05 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Heart Failure
Keywords: Cardiac Magnetic Resonance Imaging (CMR); Implantable Cardioverter Device; Implantable Loop Recorder; Left ventricular ejection fraction (LVEF); Myocardial scar
MeSH Terms: conditions — Heart Failure | interventions — Defibrillators, Implantable

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomised in a controlled fashion into two arms (n=1252):
  Arm A: ICD implantation Arm B: No ICD implantation Patients with no scar on CMR will be followed up in a registry (n=1252)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intervention (Experimental): ICD or CRTD fitted
  Interventions: Device: Implantable Cardioverter-Defibrillator (ICD) or Cardiac Resynchronisation Therapy Defibrillator (CRTD)
- Control (No Intervention): No ICD fitted (with Implantable Loop Recorder) or Cardiac Resynchronisation Therapy Pacemaker (CRTP)
- Registry (No Intervention): Usual medical care

INTERVENTIONS:
Device: Implantable Cardioverter-Defibrillator (ICD) or Cardiac Resynchronisation Therapy Defibrillator (CRTD) — An ICD is a device that is implanted under the skin under a local anesthetic. It has a battery/generator component and leads which are fixed into the heart chambers. It has the ability to detect dangerous heart rhythms if they occur, and deliver a shock to treat this to help prevent sudden cardiac death. A CRTD is a pacemaker with a defibrillator function.
  Arms: Intervention

SUMMARY:
BRITISH is a UK multicentre trial of patients who have been diagnosed with heart failure due to Non-Ischemic Cardiomyopathy (NICM, or heart failure that is not caused by blocked heart arteries. Participants will be randomised into two groups. Half the participants will receive an Implantable Cardioverter-Defibrillator (ICD) and the other half will not. The aim of the study will be to compare all-cause mortality (death from any cause) between these two groups at 36 months, and longer-term to 10 years. The study has the potential to change international heart failure treatment guidelines and to improve how patients with this condition are managed.

DETAILED DESCRIPTION:
Patients with Non-Ischemic Cardiomyopathy (NICM) have a higher risk of experiencing serious abnormal heart rhythms that might be life-threatening. Current guidelines recommend fitting a device that can correct these serious heart rhythms (Implantable Cardioverter-Defibrillator (ICD)). However, research studies have shown that 90% of patients who have an ICD will never use it because they won't experience any serious heart rhythms. A recent large trial (DANISH) of over one thousand patients with severe Non-Ischemic Cardiomyopathy has called the current guidelines into question. The trial concluded that for patients who received an ICD, there was no difference in the likelihood of dying when compared to patients that didn't have an ICD fitted. As a result, many doctors are choosing not to implant an ICD in patients with this type of heart failure, as they believe there is no overall survival benefit. However, there are clues that some patients with NICM may still benefit from an ICD, even though the headline results suggest they are not necessary. It's likely that it's the patients who are at increased risk of having a serious abnormal heart rhythm that stand to benefit from ICDs. But having an ICD fitted carries with it a significant risk of problems developing e.g. bleeding, infection, lead problems, and inappropriate shocks. These risks may not outweigh the benefits and it is this question which BRITISH will address. The study will randomly assign (like the toss of a coin), half the study participants to receive an ICD and the other half to no ICD.

Both groups will be followed up to decide whether having an ICD fitted reduces the chances of dying.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of NICM on contrast-enhanced cardiovascular magnetic resonance imaging
2. LV scar on routine CMR (patient without scar can enter the registry)
3. New York Heart Association (NYHA) Heart Failure (HF) functional class I-III and severely impaired left ventricular function (LVEF ≤ 35% on any imaging modality) after a minimum of 3 months of treatment with optimal medical therapy (OMT) as recommended by National Institute for Health and Care Excellence (NICE)
4. Able and willing to provide informed consent

Exclusion Criteria:

1. New York Heart Association (NYHA) HF functional class IV after 3 months of optimal medical therapy (OMT)
2. Acute decompensated heart failure
3. Previous implantable device in situ (PPM, Cardiac Resynchronisation Therapy (CRT) or ICD)
4. Ischemic cardiomyopathy (ICM) is defined as segmental wall motion abnormalities or wall thinning in a particular coronary territory with subendocardial or transmural late gadolinium enhancement (LGE). Patients with an LVEF ≤35% and a small amount of ischemic LGE (i.e. an infarct out of keeping with the amount of LV dysfunction) will not be excluded (so-called dual pathology patients)
5. Known diagnosis of amyloidosis, sarcoidosis, arrhythmogenic right ventricular cardiomyopathy, or hypertrophic cardiomyopathy (diseases in which there are specific guidelines regarding defibrillator therapy)
6. Known Lamin gene mutation or a positive family history of a Lamin gene mutation
7. Valve disease is considered likely to require surgery during the 3 years follow-up period
8. Complex congenital heart disease
9. Any secondary prevention ICD indication
10. Heart transplant recipient or admitted for cardiac transplantation/ left ventricular assist device
11. Clinically apparent myocardial ischemia which requires revascularization
12. Intracardiac mass which requires surgery
13. Active endocarditis
14. Active Septicaemia
15. Pregnancy
16. Life expectancy <2 years secondary to any other cause (i.e. malignancy)
17. Active treatment with chemotherapy
18. Severe renal failure (GFR <30)
19. Actively participating in another study without prior agreement between both Chief Investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2504 (Estimated)
Dates: Start 2023-04-12 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2036-04-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients alive | 3 years
  All-cause mortality

SECONDARY OUTCOMES:
Change in health-related quality of life measured using KCCQ-12 | 3 years
  Short questionnaire including questions related to heart failure symptoms and how they affect daily activities
Change in health-related quality of life measured using EQ-5D-5L | 3 years
  Questionnaire consisting of 5 questions to evaluate a patients quality of life
Cardiovascular Death | 3 years
  Percentage of patients that have cardiovascular death
Sudden cardiac death | 3 years
  Percentage of patients that have sudden cardiac death
Aborted sudden cardiac death | 3 years
  Percentage of patients that have aborted sudden cardiac death
Appropriate ICD Therapy | 3 years
  Percentage of patients that have appropriate ICD therapy
Inappropriate ICD Therapy | 3 years
  Percentage of patients that have inappropriate ICD therapy
Significant ventricular arrhythmias | 3 years
  Percentage of patients that have significant ventricular arrhythmias
NYHA Status | 3 years
  Percentage of patients in each category
Heart failure hospitalisations | 3 years
  Number of events
Cardiac hospitalisations | 3 years
  Number of events
Procedures related to implanted device | 3 years
  Number of events
Percentage of patients alive | At 5 and 10 years
  Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Flett, Study Chair — University Hospital Southampton NHS Foundation Trust
Locations (47):
- United Kingdom (47):
  - Wycombe Hospital, High Wycombe, Buckinghamshire
  - Derriford Hospital, Plymouth, Devon
  - Royal Bournemouth Hospital, Bournemouth, Dorset
  - Durham & Darlington NHS Foundation Trust, Darlington, Durham
  - Royal Sussex County Hospital, Brighton, East Sussex
  - Essex Cardiothoracic Centre, Basildon, Essex
  - James Paget University Hospitals NHS FT, Gorleston-on-Sea, Great Yarmouth
  - Portsmouth Hospitals University NHS Trust, Portsmouth, Hampshire
  - Southampton Clinical Trials Unit, Southampton, Hampshire
  - University Hospital Southampton NHS Foundation Trust, Southampton, Hampshire
  - Kent & Canterbury Hospital, Canterbury, Kent
  - Maidstone Hospital, Maidstone & Tunbridge Wells NHS Trust, Maidstone, Kent
  - Blackpool Victoria Hospiatal, Blackpool, Lancashire
  - Liverpool Heart & Chest, Liverpool, Lancashire
  - Glenfield Hospital, Leicester, Leicestershire
  - St Bartholomew's Hospital, London, London
  - Royal Free Hospital, London, London
  - Guy's Hospital, London, London
  - King's College Hospital, London, London
  - Royal Brompton Hospital, London, London
  - Hammersmith Hospital, Imperial College Healthcare NHS Trust, London, London
  - St George's Hospital, Tooting, London
  - Fairfield General Hospital, Northern Care Alliance NHS FT, Manchester, Manchester
  - Newcastle Freeman Hospital, Newcastle, Newcastle upon Tyne
  - The James Cook University Hospital, Middlesbrough, North Yorkshire
  - Wansbeck General Hospital, Ashington, Northumbria
  - Scarborough Hospital, Scarborough, Nortrh Yorkshire
  - Nottingham City Hospital, Nottingham, Nottinghamshire
  - The John Radcliffe Hospital, Oxford, Oxfordshire
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Royal Infirmary of Edinburgh, Edinburgh, Scotland
  - Musgrove Park Hospital, Taunton, Somerset
  - Northern General Hospital, Sheffield, South Yorkshire
  - University Hospital of North Tees, Hardwick, Stockton-on-Tees
  - Frimley Park Hospital, Camberley, Surrey
  - Surrey & Sussex Healthcare NHS Trust, Redhill, Surrey
  - University Hospital of Wales, Cardiff, Wales
  - University Hospital Coventry, Coventry, Warwickshire
  - New Cross Hospital, Wolverhampton, West Midlands
  - St Richards Hospital, Chichester, West Sussex
  - Leeds General Infirmary, Leeds, West Yorkshire
  - Pinderfields Hospital, Wakefield, West Yorkshire
  - Worcestershire Royal Hospital, Worcester, Worcestershire
  - Wythenshaw Hospital, Manchester, Wythenshaw
  - Castle Hill Hospital, Hull, Yorkshire
  - Royal Devon & Exeter Hospital, Exeter
  - Morriston Hospital, Swansea

IPD SHARING:
Plan to Share IPD: No